CLINICAL TRIAL: NCT06600386
Title: The Influence of Individualized Intraoperative PEEP After Alveolar Recruitment Maneuvres on the Incidence of Postoperative Respiratory Complications Following Laparoscopic Abdominal Surgery. A Prospective Randomized Controlled Study
Brief Title: Individualized Intraoperative PEEP Following Alveolar Recruitment Maneuvres and Postoperative Respiratory Complications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Collaborators: Ioanna Pikasi (Unknown)
Responsible Party: Principal Investigator, Alexandros Makris, Senior Consultant Anesthesiologist, Asklepieion Voulas General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10542/22-05-2024/AP51
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Respiratory Complications
Keywords: Alveolar Recruitment; Laparoscopy; Indvidualized PEEP

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-PEEP (Active Comparator): PEEP is standard (5cmH2O)
  Interventions: Other: Standard PEEP
- I-PEEP (Active Comparator): PEEP is individualized following standard recruitment maneuvres
  Interventions: Other: Alveolar recruitement

INTERVENTIONS:
Other: Alveolar recruitement — PEEP after alveolar reruitment maneuvres
  Arms: I-PEEP
Other: Standard PEEP — PEEP 5 cmH2O
  Arms: C-PEEP

SUMMARY:
Patients ASA I-III, undergoing laparoscopic abdominal surgery will be randomly assigned, into one of two groups, namely group C-PEEP , that will be the control group ; and group I-PEEP, where alveolar recruitment maneuvres will take place in order to identify each patient's individualized optimal PEEP. All patients will receive a standardized anesthesia regimen. The lung ultrasound score will be evaluated in all patients in the PACU and then respiratory complications will be recorded on the 24th hour, 48th hour, 7th day and 30the day, postoperatively.

ELIGIBILITY:
Inclusion Criteria:

ASA I-III Laparoscopic abdominal surgery

Exclusion Criteria:

Severe kidney dysfunction Severe hepatic dysfunction Severe respiratory disease Severe cardiac disease Severe neuromuscular disease BMI>30 Severe intraoperative hemorrage Severe intraoperative hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Respiratory complications | 30 days
  Postoperative complications (atelectasis, bronchospasm, pneumonia, respiratory failure, ARDS, prolonged mechanical ventilations, reintubation, pleural infusion, COPD exacerbation)

SECONDARY OUTCOMES:
Pplat | intraoperatively
SpO2 | intraoperatively
PCO2 | intraoperatively
PaO2/FiO2 | intraoperatively
Cdyn | intraoperatively
Ppeak | intraoperatively
MAP | intraoperatively
heart rate | intraoperatively
LUS score | Preoperatively and 30 minutes postoperatively
  Ultrasonographic findigs

CONTACTS AND LOCATIONS:
Locations (1):
- Asklepieion Hospital of Voula, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided